CLINICAL TRIAL: NCT04616625
Title: Cardiovascular Effects of Prenatal Methamphetamine Exposure
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Adventist Health and Rideout (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1632548
Record Dates: First submitted 2020-10-08; First posted 2020-11-05 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Methamphetamine Abuse; Newborn Complication | Patient | Neonatalology
Keywords: Methamphetamine; Methamphetamine in pregnancy; Cardiovascular effects of methamphetamine on newborn; Effect of prenatal methamphetamine exposure on neurodevelopment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methamphetamine exposed: Infants born to mothers with prenatal history of MA use during current pregnancy and/or positive meconium toxicology positive for MA in infant.
- Methamphetamine non-exposed: Infants born to mothers without prenatal history of MA use during this pregnancy and negative meconium toxicology for MA in infant.

SUMMARY:
Methamphetamine (MA) is one of the commonly used drugs during pregnancy. Cardiovascular effects of MA include elevated blood pressure, acute vasospasm, atherosclerotic disease, structural and electrical remodeling of cardiac tissue leading to arrhythmias and heart failure, and pulmonary hypertension.1 In addition, MA can cause neurotoxicity with harmful effects on neurodevelopment in the children who had prenatal exposure.5-8 Currently neonatal providers do not perform detailed cardiovascular evaluation in newborn period or long term neurodevelopmental assessments as outpatient for the newly born infants with prenatal exposure to MA, and they do not qualify for early intervention. The goal of the investigators is to perform detailed cardiovascular evaluation in neonatal period and estimate baseline prevalences and follow up with developmental and cardiovascular assessment using a questionnaire at 12 months in a cohort of neonates enriched with those who had prenatal exposure to MA.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born at UCDCH and at AHRO at gestational age >34 weeks. (<34 weeks excluded to avoid the effects of prematurity)
2. For the MA exposed subgroup (n=30): Infants born to mothers with prenatal history of MA use during current pregnancy and/or positive meconium toxicology positive for MA in infant.
3. For the MA unexposed subgroup (n=12): Infants born to mothers without prenatal history of MA use during this pregnancy and negative meconium toxicology for MA in infant.

Exclusion Criteria:

a) Presence of congenital anomalies and known fatal conditions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants born at UCDCH and at AHRO at gestational age >34 weeks. (<34 weeks excluded to avoid the effects of prematurity)
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Estimation of prevalence of MA use among births | Through study completion, an average of 2 years.
Evaluation of effects of prenatal MA exposure on neonatal cardiovascular status. | Through study completion, an average of 2 years.
  Perfusion index by pulse-oximeter, heart function by echocardiogram, EKG and detailed cardiac exam in the newborn period between 24-48 hours after birth.

SECONDARY OUTCOMES:
Infant's neurodevelopmental outcome and general assessment at 12 months of age. | Through study completion, an average of 2 years.
  Phone call with parent to assess the infant's neurodevelopment at 12 months of age using "Ages and Stages" questionnaire with parent and/or pediatrician, assessment of general health, nutrition and cardiovascular status (BP measurement) by phone call with pediatrician

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Adventist Health and Rideout, Marysville, California
  - UC Davis Children's Hospital, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/cardiovascular-effects-of-prenatal-methamphetamine-exposure-546096/